CLINICAL TRIAL: NCT05540847
Title: Comparison of Interfascial Injection Versus Subpectineal Injection on Ultrasound-guided Obturator Nerve Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Halil Cihan Kose, Principal investigator, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 141/09
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Bladder Neoplasm
Keywords: obturator nerve block; ultrasound guided block; bladder tumor
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound guided interfascial obturator nerve block (Active Comparator): In supine position, ultrasound probe will be placed on inguinal region, 2-3 cm below to the inguinal crease. Patients in this group will receive interfascial obturator nerve block under ultrasound guidance.
  Interventions: Procedure: Interfascial Injection
- Ultrasound guided subpectineal obturator nerve block (Experimental): In supine position, the ultrasound probe will be placed on in inguinal region, 1-2 cm below to the inguinal crease to identiy the subpectineal area. Patients in this group will receive subpectineal obturator nerve block under ultrasound guidance.
  Interventions: Procedure: Subpectineal Injection

INTERVENTIONS:
Procedure: Interfascial Injection — Interfascial Injection on Ultrasound-guided Obturator Nerve Block
  Arms: Ultrasound guided interfascial obturator nerve block
Procedure: Subpectineal Injection — Subpectineal Injection on Ultrasound-guided Obturator Nerve Block
  Arms: Ultrasound guided subpectineal obturator nerve block

SUMMARY:
This study aimed to assess the effectiveness of the ultrasound-guided interfascial injection approach with the subpectineal injection technique for obturator nerve block in bladder cancers undergoing transurethral resection of bladder tumor (TURBT) under spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Lateral wall bladder tumour
* ASA I-II patients

Exclusion Criteria:

* Contraindications for spinal anesthesia,
* Tumors that disrupt the integrity of the bladder,
* Coagulation disorders,
* Uncooperative patients,
* Allergy to local anesthetics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-16 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-23 (Actual)

PRIMARY OUTCOMES:
Success rate of obturatr nerve block | Peroperative period
  The success or fail of the obturator nerve block will be conformed using nerve stimulator. Detecting muscles twitch will br considered to be a fail.

SECONDARY OUTCOMES:
Number of adductor muscle spazms | Intraoperative period
  Number of adductor muscle spazms in each group will be noted during the intraoperative period.
Sensory block | 30 minutes after the intervention
  Sensory block area will be evaluated by a pin prick at in the dermatomal areas related obturator nerve and branches.
Patient satisfaction | Peroperative period
  Changes in overall satisfaction will be assessed using a 5 point Likert Scale ( 1-very dissatisfied, 2- dissatisfied, 3- neutral, 4-satisfied, 5 - very satisfied
Procedure time | During the procedure
  Block performance time will be recorded from the time the first ultrasound image is obtained until the procedure is completed

CONTACTS AND LOCATIONS:
Locations (1):
- Health Science University Diskapi Yildirim Beyazıt Training and Research Hospital, Yenimahalle, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No